CLINICAL TRIAL: NCT01583777
Title: A Phase 1 Study for the Evaluation of Excretion (Mass Balance) and Pharmacokinetics of 14C-Labeled Belinostat in Patients With Advanced Cancer
Brief Title: Phase I Mass Balance, PK and Safety Study of 14C-Labeled Belinostat in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acrotech Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPI-BEL-12-103
Record Dates: First submitted 2012-04-19; First posted 2012-04-24 (Estimated); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Advanced Cancer
Keywords: Belinostat
MeSH Terms: interventions — belinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Belinostat (Experimental): Open Label
  Interventions: Drug: Belinostat

INTERVENTIONS:
Drug: Belinostat — On Day 1, a single dose of 14C-labeled belinostat (approximately 94 to 105 µCi, 1500 mg) will be administered to the patient as a 30-minute IV infusion.
  After Cycle 1 evaluations are completed, and if it is in the best interest of the patient, patients may receive additional cycles of non-radiolabeled belinostat until disease progression, unacceptable toxicity, or initiation of new anticancer therapy. After Cycle 1, Day 21, non radiolabeled belinostat will be administered IV as a 30 -45 minute infusion of 1000 mg/m2 on Days 1 through 5 every 21 days.
  Other Names: beleodaq

SUMMARY:
The purpose of this trial is to study the mass balance, pharmacokinetics (PK), and safety of belinostat following IV administration in patients with a recurrent or progressive malignancy.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, single-dose study of 14C-labeled belinostat to determine routes of elimination of belinostat. A single dose of 14C-labeled belinostat (approximately 94.3 to 105 µCi, 1500 mg) will be administered as a 30-minute IV infusion to the patient. Routes of elimination of belinostat and its metabolites will be assessed by estimating the recovery of total radioactivity and parent belinostat over a period of 7 days. Plasma samples will be taken for 3 days at specified intervals for PK assessments. Total radioactivity in plasma, urine, and feces will be determined by liquid scintillation counting. Concentrations of belinostat in plasma and urine will be determined using a validated liquid chromatography - tandem mass spectroscopy (LC-MS/MS) method. Selected plasma, urine, and feces samples will be retained for use in the metabolism investigation. Samples will be initially analyzed using radio-high performance liquid chromatography (HPLC) to determine the number and relative proportion of belinostat and metabolites present. Selected samples will be subsequently analyzed using LC-MS to identify the major metabolites (> 10% of parent area under the curve [AUC]). If it is in the interest of the patient, treatment with non-radiolabeled belinostat may be continued with 21-day cycles until disease progression, initiation of new anticancer therapy, or an adverse event (AE) that may affect patient participation.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent document indicating understanding of the purpose of and procedures required for the study and willingness to participate in the study.
2. Histological confirmation of cancer and refractory or intolerant to standard therapy or cancer for which no standard therapy exists.
3. Age at study entry of 18 years or older.
4. Availability to stay in the research unit for the first 7 days.
5. Adequate renal function defined as a calculated creatinine clearance (CrCl) of > 45 mL/minute.
6. Adequate hepatic function: total bilirubin < 1.5 x the upper limits of normal (ULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 x ULN.
7. Adequate hematopoietic function defined as an absolute neutrophil count (ANC) > 1000 cells/µL and platelet count > 50,000/µL.
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
9. Life expectancy of at least 12 weeks.
10. If female, patient must be postmenopausal for at least 1 year, documented surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy), or of childbearing potential and practicing birth control. Acceptable contraceptive methods in this study are intrauterine device; diaphragm or condom in combination with spermicidal foam or jelly; injectable, implantable, or transdermal patch; or oral contraception.
11. Female patients must have a negative pregnancy test at the Screening Visit and at the end of study treatment (30 days after the last dose of belinostat).

Exclusion Criteria:

1. Known anal or urinary incontinence.
2. Diagnosis of acute myelogenous leukemia (AML), multiple myeloma, primary hepatic or renal carcinomas.
3. Inability to consume oral fluids.
4. Treatment with drugs known to inhibit metabolic pathways (glucuronidation, CYP system) in the 4 weeks before the Screening Visit.
5. Concurrent treatment with diuretics or laxatives.
6. Radiotherapy involving mouth, esophagus, and gastrointestinal tract in the 4 weeks before the Screening Visit.
7. Polymorphism in UGT1A1.
8. Known diagnosis of human immunodeficiency virus (HIV), hepatitis B or C.
9. Previous participation in a study utilizing 14C.
10. Body surface area < 1.5 m2.
11. Ongoing or medical history of a physical or psychiatric illness, significant comorbidity, or any medical disorder other than cancer that may require treatment or make the subject unlikely to fully complete the study.
12. Use of another investigational product or anticancer agent within 4 weeks prior to the Screening Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Maximum recovery of the radioactive dose in urine and feces | 6 months
  The route of elimination of belinostat will be determined by the recovery of total radioactivity (parent drug and metabolites) and unmetabolized belinostat in urine and feces following single IV administration of 14C-labeled belinostat in patients with recurrent or progressive malignancy.

SECONDARY OUTCOMES:
The Concentration of Belinostat in plasma, urine, and feces and its metabolites | 6 months
  Secondary objectives are to determine the PK of 14C-labeled belinostat in plasma, urine, and feces following IV administration; to determine the relative proportion of 14C-labeled belinostat and its radiolabeled metabolites in plasma, urine, and feces; and to assess the safety of belinostat.

CONTACTS AND LOCATIONS:
Overall Officials: Mi R Choi, MD, Study Director — Spectrum Pharmaceuticals, Inc
Locations (1):
- Hospital Universitario Madrid Sanchinarro, Madrid, Spain